CLINICAL TRIAL: NCT02259192
Title: Cochlear Implantation for Single-Sided Deafness
Brief Title: Cochlear Implants for Adults With Single-sided Deafness
Acronym: SSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Robert Shannon (Other)
Collaborators: Med-El Corporation (Industry); House Clinic, Inc. (Industry); University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Robert Shannon, Professor of Research, Otolaryngology - Head and Neck Surgery, University of Southern California
Organization: University of Southern California (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CI for SSD adults
Record Dates: First submitted 2014-09-26; First posted 2014-10-08 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Single-sided Deafness
Keywords: deaf adult; single-sided; cochlear implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label (Experimental): Cochlear Implant
  Interventions: Device: MED-EL Maestro Cochlear Implant

INTERVENTIONS:
Device: MED-EL Maestro Cochlear Implant — cochlear implant

SUMMARY:
The purpose of this investigation is to determine the safety and preliminary efficacy of implanting a cochlear implant (CI) in the profoundly deaf ear of an adult with one normal hearing (NH) ear (termed "single-sided deaf" person, or SSD). The potential subjects will have been deafened post-lingually, thus, at one point the now deafened ear did conduct sound from the periphery. The MED-EL CI system will be implanted in ten (10) SSD patients.The long-term goal of this research program is to determine whether the CI, in combination with the NH ear, may provide improved localization ability and better speech understanding in noise, relative to performance before cochlear implantation (i.e., with the NH ear alone). A secondary long-term goal is to determine whether CI stimulation may reduce tinnitus severity, compared to tinnitus experienced prior to cochlear implantation or when the CI is turned off, after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Is an adult (18 years of age or older)
* English as the primary language
* Able to undergo general anesthesia, as determined by physical examination and written report from the physician
* Receives pneumovax vaccine within 2 weeks of surgery and provides documentation to the principal investigator
* Profoundly/severely deaf in one ear ("implant ear"), as defined by:

  * 3-frequency pure-tone average≥70 dB Hearing Loss
  * Bone conduction thresholds consistent with air conduction thresholds (i.e., no conductive component to the hearing loss)
  * HINT sentence recognition score ≤40% correct, 60 dBA presentation level
  * Post-lingual onset of hearing loss, i.e., after age 6 years of age
  * Hearing loss occurred <10 years prior, as obtained by history
* Normal hearing in one ear ("non-implant ear"), as defined by:

  * 3-frequency PTA ≤25 dB HL
  * No tested frequency air conduction threshold >35 dB HL
  * Bone conduction thresholds consistent with air conduction thresholds
  * Word recognition score ≥80% correct, 60 dBA presentation level
  * HINT sentence recognition score ≥ 80%, 60 dBA presentation level
* Provides informed consent
* Willing and able to follow the study protocol

Exclusion Criteria:

* Retrocochlear pathology resulting from Neurofibromatosis 2, or other types of cranial nerve/brainstem tumors
* Co-existing medical conditions that require radiotherapy of the brainstem and/or auditory cortex
* Any medical contraindication precluding safe administration of general anesthesia, e.g.,

  * Cardiopulmonary disease
  * Renal disease
* Otologic conditions which contraindicate surgery

  * Active middle ear infection
  * Tympanic membrane perforation
* Anatomic abnormalities detected on CT preventing appropriate placement of the stimulator housing in the bone of the skull or placement of the electrode array in the cochlea (e.g., ossification)
* Psychological conditions contraindicating surgery
* Skin or scalp conditions that may preclude attachment of the coil or that may interfere with the use of the coil
* Chronic pain in or around the head
* Current or previous use of an active hearing implant (e.g., bone-anchored hearing aids, cochlear implant, etc.)
* Developmental delays or organic brain dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Pure-tone threshold average (dB) | 6 months post-activation
  Change in 3-frequency pure-tone threshold average (dB) in the normal hearing ear.
Hearing in Noise Test (signal-to-noise ratio) | 6 months post-activation
  Change in Hearing in Noise Test signal-to-noise ratio in the normal hearing ear.

SECONDARY OUTCOMES:
Adverse Events | 1-month post-implantation
  Number of unexpected serious adverse events across all 10 subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shannon, PhD, Principal Investigator — Keck School of Medicine of USC
Locations (2):
- United States (2):
  - Keck School of Medicine of USC, Los Angeles, California
  - House Clinic, Los Angeles, California